CLINICAL TRIAL: NCT06741449
Title: The Outcomes of Keystone Perforator Island Flap Versus Lay Open in Re-recurrent Pilonidal Sinus Disease ( Two Times of Recurrence or More): One Year Experience Study
Brief Title: The Outcomes of Keystone Perforator Island Flap Versus Lay Open in Re-recurrent Pilonidal Sinus Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, lecturer of general surgery, faculty of medicine, Zagazig University, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #881\8-Dec-2024
Record Dates: First submitted 2024-12-09; First posted 2024-12-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-12

CONDITIONS: Pilonidal Sinus Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- re- recurrent pilonidal sinus (Active Comparator)
  Interventions: Procedure: keystone flap
- re-recurrent pilonidal sinus (Active Comparator)
  Interventions: Procedure: lay open

INTERVENTIONS:
Procedure: keystone flap — facio-cutaneous flap used to cover the defect after removal of the disease
  Arms: re- recurrent pilonidal sinus
Procedure: lay open — after removal of the disease, the wound is left open to heal by granulation tissue
  Arms: re-recurrent pilonidal sinus

SUMMARY:
Pilonidal disease is a common and annoying problem with a fair recurrence rate. Every time of recurrence more skin is needed to cover the defect and if left open healing is supposed to be prolonged.

ELIGIBILITY:
Inclusion Criteria:

* re-recurrent pilonidal disease

Exclusion Criteria:

* patients with proved anal or perineal malignancy or autoimmune disease
* patient with pilonidal disease for the first time or for the first time of recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
operative time | operative time is measured in minutes from incision to wound dressing
bleeding amount | amount of blood lost is measured from incision for 2 days post operative
  intra and post operative bleeding amount is measured in cc by volumetric method
healing time | healing time is measured for 3 months post-operatively
wound infection | wound infection is evaluated for 3 months post-operatively
  wound infection evaluated by presence of pus from the first day post-operativel

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
data will be available on demand by contacting the principle investigator